CLINICAL TRIAL: NCT05404230
Title: Prevention of Oxaliplatin-induced Peripheral Neuropathy - a Randomized Controlled Trial
Brief Title: Prevention of Oxaliplatin-induced Nerve Damage in the Body's Extremities
Acronym: OxaNeuro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OxaNeuro
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Neuropathy; Colorectal Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Colorectal Neoplasms | interventions — Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil (Active Comparator): 4 capsules containing n-3 poly unsaturated fatty acids (EPA and DHA) with a total concentration of 3 g per day.
  4 capsules per day for 8 months
  Interventions: Dietary Supplement: Fish oil
- Corn oil (Placebo Comparator): 4 capsules containing n-6 poly unsaturated fatty acids in a total concentration of 2 g per day.
  4 capsules per day for 8 months.
  Corn oil is regularly used in the kitchen and the daily dose in the study is the equivalent of adding an extra spoon of food oil when cooking. It has no known effect on the parameters we want to examine.
  Interventions: Dietary Supplement: Corn oil

INTERVENTIONS:
Dietary Supplement: Fish oil — Fish oil containing poly unsaturated fatty acids.
  Arms: Fish oil
Dietary Supplement: Corn oil — Corn oil
  Arms: Corn oil

SUMMARY:
The purpose of this study is to examine the effect of supplementary polyunsaturated fatty acids on nerve damage in the body's extremitites of patients treated with oxaliplatin containing chemotherapy after surgery for colorectal cancer.

DETAILED DESCRIPTION:
The primary objective of the present study is to examine if a high dosage of n-3 PUFA reduces the incidence and severity of chemotherapy-induced peripheral neuropathy (CIPN) 8 months after adjuvant oxaliplatin following surgery for high-risk colorectal cancer.

An additional aim is to investigate whether n-3 PUFAs have an effect on nutritional status, cognition and mental status. Inflammatory mechanisms and biomarkers of CIPN in skin biopsies and in blood will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified adenocarcinoma of the colon or rectum and planned standard adjuvant treatment with capecitabine in combination with oxaliplatin.
* ECOG performance status 0-2 (measurement of a patient's function in terms of self-care, daily activity and physical ability.
* Written and orally informed informed consent

Exclusion Criteria:

* Inability to speak, read, and understand Danish.
* Previous treatment with neurotoxic chemotherapy.
* Neurological (including neuropathy) or psychiatric disorders, diabetes or other significant medical conditions.
* Alcohol or drug abuse.
* Sensory disturbances in the feet
* Spinal stenosis.
* Vascular disease (Fontaine grade II or more).
* Known allergy to fish, fish oil or corn oil
* Fertile patients not willing to use effective methods of contraception during treatment or abstinence.
* Daily intake of oil supplements and not willing to stop during the trial period.
* Lack of consent to skin biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced peripheral neuropathy (CIPN) 8 months after start of adjuvant chemotherapy | 8 months after start of adjuvant chemotherapy
  Number of patients who meet the criteria for CIPN: relevant symptoms evaluated by a medical doctor, incl one of the following: abnormal vibration test or, abnormal nerve conduction test by DPN check device or, abnormal pinprick test or, abnormal skin biopsy.

SECONDARY OUTCOMES:
Intensity of CIPN-related neuropathic pain 8 months after adjuvant chemotherapy according to the Numeric Rating Scale (NRS) | 8 months after start of adjuvant chemotherapy
  Average over the past 24 hours measured by NRS (scale from 0-10 with 0=no pain and 10=worst pain imaginable)
Change in severity of CIPN from baseline to 8 months after start of adjuvant chemotherapy according to the EORCT QLQ-CIPN 20 questionnaire | 8 months after start of adjuvant chemotherapy
  EORCT QLQ-CIPN 20 = the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Lise Ventzel, MD PHD, Study Director — medical doctor at Vejle Hospital, University Hospital of southern Denmark
Locations (1):
- Deparment of Oncology, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Due to restrictions related to Danish law protecting patient privacy, the data used in this study can be made available if it complies with GDPR and through an application to the Region of Southern Denmark
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Due to restrictions related to Danish law protecting patient privacy, the data used in this study can be made available if it complies with GDPR and through an application to the Region of Southern Denmark
Access Criteria: Due to restrictions related to Danish law protecting patient privacy, the data used in this study can be made available if it complies with GDPR and through an application to the Region of Southern Denmark

REFERENCES:
- [Derived] Gehr NL, Karlsson P, Timm S, Christensen S, Hvid CA, Peric J, Hansen TF, Lauritzen L, Finnerup NB, Ventzel L. Study protocol: fish oil supplement in prevention of oxaliplatin-induced peripheral neuropathy in adjuvant colorectal cancer patients - a randomized controlled trial. (OxaNeuro). BMC Cancer. 2024 Feb 3;24(1):168. doi: 10.1186/s12885-024-11856-z. PMID 38308227